CLINICAL TRIAL: NCT00776633
Title: Intracoronary Stenting and Antithrombotic Regimen: Testing of a Six-week Versus a Six-month Clopidogrel Treatment Regimen in Patients With Concomitant Aspirin and Oral Anticoagulant Therapy Following Drug-eluting Stenting
Brief Title: Triple Therapy in Patients on Oral Anticoagulation After Drug Eluting Stent Implantation
Acronym: ISAR-TRIPLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. A01508
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation
Keywords: aspirin; clopidogrel; oral anticoagulation; warfarin; drug eluting stent; phenprocoumon
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short triple (Experimental): 6 weeks triple therapy
  Interventions: Drug: aspirin; Drug: clopidogrel; Drug: oral anticoagulation
- Long triple (Active Comparator): 6 months triple therapy
  Interventions: Drug: aspirin; Drug: clopidogrel; Drug: oral anticoagulation

INTERVENTIONS:
Drug: aspirin — 6 weeks triple therapy with aspirin, clopidogrel and oral anticoagulation
Drug: clopidogrel — 6 months triple therapy with aspirin, clopidogrel and oral anticoagulation
Drug: oral anticoagulation

SUMMARY:
The investigators hypothesize that reducing the duration of clopidogrel therapy from 6 months to 6 weeks after DES implantation is associated with improved clinical outcomes in patients on ASA and an oral anticoagulant.

DETAILED DESCRIPTION:
The introduction of drug-eluting stents (DES) was associated not only with a widening of the indication for percutaneous coronary intervention (PCI) but also with longer antithrombotic therapy duration. Dual antiplatelet therapy with ASA and a thienopyridine is very efficient in preventing adverse events after coronary stenting but it is inferior to oral anticoagulation (OAC) to reduce the risk of stroke in patients with atrial fibrillation. OAC is also superior to antiplatelet therapy in patients with mechanical heart valves and the therapy of choice for the treatment of deep vein thrombosis and pulmonary embolism. OAC is also administered for left ventricular thrombi and low ejection fraction. There is an increasing number of patients undergoing coronary stenting who are in need of life-long anticoagulation therapy and would therefore require a triple therapy consisting of aspirin, clopidogrel and oral anticoagulation. As oral anticoagulation and antithrombotic therapy impair primary and secondary hemostasis there are concerns that adding warfarin to dual antiplatelet therapy might cause increased bleeding rates. Several studies have retrospectively assessed efficacy and safety in patients receiving a triple therapy with various results: major bleeding rates varied from 3,1%-14,9% with total bleeding rates up to 27,5%. Prospective randomized data on this topic are not available. Therefore the aim of this study is to compare a 6 week versus a 6 month triple therapy after DES implantation.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with an indication for oral anticoagulation and a DES implantation.
2. Informed, written consent by the patient or her/his legally-authorized representative for participation in the study.

Key Exclusion Criteria:

1. Age ≤18 years
2. Previous stent thrombosis
3. DES in left main

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Composite of death, myocardial infarction, definite stent thrombosis, stroke or major bleeding. | 9 months

SECONDARY OUTCOMES:
Ischemic complications (composite of cardiac death, myocardial infarction, stent thrombosis or ischemic stroke) | 9 months
Bleeding complications (Major bleeding) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentum München; Stefanie Schulz, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (3):
- Aarhus University Hospital, Aarhus, Denmark
- Germany (2):
  - Deutsches Herzzentrum München, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Background] Rubboli A, Halperin JL, Airaksinen KE, Buerke M, Eeckhout E, Freedman SB, Gershlick AH, Schlitt A, Tse HF, Verheugt FW, Lip GY. Antithrombotic therapy in patients treated with oral anticoagulation undergoing coronary artery stenting. An expert consensus document with focus on atrial fibrillation. Ann Med. 2008;40(6):428-36. doi: 10.1080/07853890802089786. PMID 18608125
- [Background] Schomig A, Neumann FJ, Kastrati A, Schuhlen H, Blasini R, Hadamitzky M, Walter H, Zitzmann-Roth EM, Richardt G, Alt E, Schmitt C, Ulm K. A randomized comparison of antiplatelet and anticoagulant therapy after the placement of coronary-artery stents. N Engl J Med. 1996 Apr 25;334(17):1084-9. doi: 10.1056/NEJM199604253341702. PMID 8598866
- [Derived] Fiedler KA, Maeng M, Mehilli J, Schulz-Schupke S, Byrne RA, Sibbing D, Hoppmann P, Schneider S, Fusaro M, Ott I, Kristensen SD, Ibrahim T, Massberg S, Schunkert H, Laugwitz KL, Kastrati A, Sarafoff N. Duration of Triple Therapy in Patients Requiring Oral Anticoagulation After Drug-Eluting Stent Implantation: The ISAR-TRIPLE Trial. J Am Coll Cardiol. 2015 Apr 28;65(16):1619-1629. doi: 10.1016/j.jacc.2015.02.050. PMID 25908066
- [Derived] Fiedler KA, Byrne RA, Schulz S, Sibbing D, Mehilli J, Ibrahim T, Maeng M, Laugwitz KL, Kastrati A, Sarafoff N. Rationale and design of The Intracoronary Stenting and Antithrombotic Regimen-Testing of a six-week versus a six-month clopidogrel treatment Regimen In Patients with concomitant aspirin and oraL anticoagulant therapy following drug-Eluting stenting (ISAR-TRIPLE) study. Am Heart J. 2014 Apr;167(4):459-465.e1. doi: 10.1016/j.ahj.2014.01.005. Epub 2014 Jan 14. PMID 24655693